CLINICAL TRIAL: NCT03198260
Title: Influence of Fascial Manipulation on Running Kinematics Among Athletes With Medial Tibial Stress Syndrome.
Brief Title: Observing the Effect of Fascial Manipulation in Athletes With Shin Splits.Tibial Stress Syndrome.
Acronym: MTSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Siddhant Shipurka, Postgraduate student, Manipal University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTRI/2017/06/008875
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Shin Splint; Fascial Manipulation; Running Kinematics
MeSH Terms: conditions — Medial Tibial Stress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial Manipulation (Experimental): fascial manipulation is a manual therapy technique were to apply deep frictional massage to the deep fascial structure or point to increase its pliability
  Interventions: Other: Fascial manipulation
- Running kinematics (Active Comparator): the change in a range of joint angles during different phases of running
  Interventions: Other: Fascial manipulation

INTERVENTIONS:
Other: Fascial manipulation — Deep frictional massage

SUMMARY:
Aims & objectives:

1. The aim of the study is to find out the influence of fascial manipulation on running kinematics among athletes with medial tibial stress syndrome (MTSS).
2. The objectives of our study are

i. To use fascial manipulation as a mode of treatment in MTSS. ii. To compare running kinematics before and after treatment intervention. iii. To compare pain perception before and after treatment intervention.

DETAILED DESCRIPTION:
The justification for study:

1. MTSS is associated with altered lower extremity kinematics.
2. There is an association between tibial fascia tightness and forces acting along the tibial crest due to alterations in the transfer of energy from foot proximally in the closed kinematic chain.
3. Fascial manipulation is found to be effective in improving the pliability of connective tissues in the management of musculoskeletal conditions.
4. Therefore there is a need to determine the influence of fascial manipulation on MTSS.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-40 years, both sexes Athletes with shin pain or diagnosed with MTSS Symptoms lasting for 2-3 weeks in the last 1 month

Exclusion Criteria:

* Trauma to lower extremity in the past 3 months Neurological, Cognitive, Psychological factors affecting the test Acute injuries- laceration, sprains, strains, recent fractures Lumbopelvic-hip complex and knee pathologies(intra-articular lesions, osteoarthritis, rheumatic arthritis, osteomyelitis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | After 5 to 10 mins
  Self reporting pain intensity after resuming running

SECONDARY OUTCOMES:
Increase in running economy | 15 mins to 45 mins
  Increasing in duration of running compared to the first trial

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sport Science Medicine and Research, Udupi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reshef N, Guelich DR. Medial tibial stress syndrome. Clin Sports Med. 2012 Apr;31(2):273-90. doi: 10.1016/j.csm.2011.09.008. PMID 22341017
- [Result] Winkelmann ZK, Anderson D, Games KE, Eberman LE. Risk Factors for Medial Tibial Stress Syndrome in Active Individuals: An Evidence-Based Review. J Athl Train. 2016 Dec;51(12):1049-1052. doi: 10.4085/1062-6050-51.12.13. Epub 2016 Nov 11. PMID 27835043
- [Result] Newman P, Witchalls J, Waddington G, Adams R. Risk factors associated with medial tibial stress syndrome in runners: a systematic review and meta-analysis. Open Access J Sports Med. 2013 Nov 13;4:229-41. doi: 10.2147/OAJSM.S39331. PMID 24379729
- [Result] Brown AA. Medial Tibial Stress Syndrome: Muscles Located at the Site of Pain. Scientifica (Cairo). 2016;2016:7097489. doi: 10.1155/2016/7097489. Epub 2016 Mar 15. PMID 27066291
- [Result] Souza RB. An Evidence-Based Videotaped Running Biomechanics Analysis. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):217-36. doi: 10.1016/j.pmr.2015.08.006. Epub 2015 Oct 20. PMID 26616185
- [Result] Winters M, Eskes M, Weir A, Moen MH, Backx FJ, Bakker EW. Treatment of medial tibial stress syndrome: a systematic review. Sports Med. 2013 Dec;43(12):1315-33. doi: 10.1007/s40279-013-0087-0. PMID 23979968
- [Result] Mikolajczyk A, Kociecki M, Zaklukiewicz A, Listewnik M, Gebska M. [USE OF THE STRUCTURAL TENSEGRATION CONCEPT IN THE STECCO FASCIAL MANIPULATION METHOD]. Ann Acad Med Stetin. 2014;60(2):59-64. Polish. PMID 26591110
- [Result] Stecco C, Day JA. The fascial manipulation technique and its biomechanical model: a guide to the human fascial system. Int J Ther Massage Bodywork. 2010 Mar 17;3(1):38-40. doi: 10.3822/ijtmb.v3i1.78. No abstract available. PMID 21589701